CLINICAL TRIAL: NCT00718562
Title: A Multi-center Phase II Study to Evaluate the Efficacy and Safety of AMN107 (Nilotinib) in Patients With Gastrointestinal Stromal Tumors Who Have Progressed on or Are Intolerant to Both Imatinib and Sunitinib
Brief Title: Efficacy and Safety of AMN107 in Patients With GastroIntestinal Stromal Tumors (GIST) Who Have Failed Both Imatinib and Sunitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107D1201
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: nilotinib; AMN107; Sunitinib; Sunitinib malate; Imatinib; Imatinib mesylate; Tyrosine
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: AMN107

INTERVENTIONS:
Drug: AMN107

SUMMARY:
This study will evaluate the efficacy and safety of nilotinib in gastrointestinal stromal tumors patients who failed imatinib and sunitinib therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented disease progression during imatinib and sunitinib therapy OR intolerance to imatinib and/or sunitinib
* At least one measurable site of disease on CT/MRI scan
* PS≤2
* Normal organ, electrolyte, and bone marrow function

Exclusion Criteria:

* Previous treatment with nilotinib or any other drug in this class or other targeted therapy
* Treatment with any cytotoxic and/or investigational drug ≤ 4 weeks prior to study entry
* Impaired cardiac function
* Use of coumarin derivatives (i.e. warfarin)
* Women who are pregnant or lactating

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) in all patients with either sunitinib-resistant GIST or in patients with GIST who are intolerant of sunitinib | 24 weeks

SECONDARY OUTCOMES:
DCR in patients with sunitinib-resistant GIST, Progression free survival (PFS), overall survival (OS), Objective response rate (ORR) | 24 weeks
Safety | 24 weeks
PK profile | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Japan (8):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Niigata, Niigata
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Sunto-gun, Shizuoka
  - Novartis Investigative Site, Chuo-ku, Tokyo

REFERENCES:
- [Result] Sawaki A, Nishida T, Doi T, Yamada Y, Komatsu Y, Kanda T, Kakeji Y, Onozawa Y, Yamasaki M, Ohtsu A. Phase 2 study of nilotinib as third-line therapy for patients with gastrointestinal stromal tumor. Cancer. 2011 Oct 15;117(20):4633-41. doi: 10.1002/cncr.26120. Epub 2011 Mar 31. PMID 21456006